CLINICAL TRIAL: NCT01632358
Title: A Randomized, Double-blind, Placebo Controlled, Crossover Study to Assess Safety and Tolerability, Pharmacokinetics, and Explore Pharmacodynamics of TAP311 in Patients With Mixed Dyslipidaemia
Brief Title: Safety and Pharmacokinetis of TAP311 in Dyslipidemic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTAP311X2201; 2012-000857-29
Record Dates: First submitted 2012-06-28; First posted 2012-07-02 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Dyslipidaemia
Keywords: safety; tolerability; pharmacokinetics
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP311 capsules (Experimental): Patients will receive TAP311 capsule orally once daily for 14 days.
  Interventions: Drug: TAP311 capsules
- Placebo of TAP311 capsules (Placebo Comparator): Matching placebo to TAP311 capsule, once daily for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAP311 capsules
  Arms: TAP311 capsules
Drug: Placebo
  Arms: Placebo of TAP311 capsules

SUMMARY:
The study will assess the safety, tolerability and pharmacokinetics of TAP311 in patients with dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 to 80 years (inclusive) of age.
* Patients are not treated for dyslipidemia with medications other than HMG-CoA reductase inhibitors (statins) for at least 4 weeks prior to Day 1. Patients should be on stable doses of current medications, if any, for at least 3 months to be eligible.
* Patients must weigh at least 50 kg to participate in the study, and must have a body mass index (BMI) within the range of 18 - 40 kg/m2.

Exclusion Criteria:

* Use of other investigational drugs at the time of enrollment
* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes
* Use of lipid modifying agents (e.g. fenofibrate, niacin, omega-3 fatty acids, etc.) other than statins will exclude subjects.
* Pregnant or nursing (lactating) women
* Diabetic patients whose plasma glucose is not well controlled by stable diabetic treatment for at least 3 months
* Heavy smokers (smoke more than 10 cigarettes a day routinely and who cannot refrain from smoking during the study).
* Women of child-bearing potential (WOCBP) can be included but must use highly effective contraception
* Significant illness within two (2) weeks prior to initial dosing
* History of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result.
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | 14 days after treatment
  Summary statistics on number of patients with total adverse events, serious adverse events and death will be reported.

SECONDARY OUTCOMES:
Pharmacokinetics of TAP311: The observed maximum plasma concentration following drug administration at steady state (Cmax,ss) | Day 1 and Day 14
  Day 1 - Cmax, Day 14 - Cmaxss, from the plasma concentration-time data. Each parameters will be one outcome measure
Pharmacokinetics of TAP311: The time to reach the maximum concentration after drug administration at steady state(Tmax, ss) | Day 1 and Day 14 profile
  The time to reach the maximum concentration after drug administration at steady state(Tmax, ss)
Pharmacokinetics of TAP311: The area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) | Day 1
  The area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast)
Pharmacokinetics of TAP311: The Racc ratio from the plasma concentration-time data | Day 14
  The Racc ratio from the plasma concentration-time data
Pharmacokinetics of TAP311: The AUCtau, from the plasma concentration-time data | Day 14
  The AUCtau, from the plasma concentration-time data

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Novartis Investigative Site, Miramar, Florida, United States
- Novartis Investigative Site, Amman, Jordan
- Novartis Investigative Site, Taichung, Taiwan, Taiwan